CLINICAL TRIAL: NCT02955368
Title: A Multi-center, Randomized, Double-blind, Parallel-group Phase III Clinical Trial to Evaluate the Efficacy and Safety of DP-R212 Fixed Dose Combination in Patients With Dyslipidemia and Hypertension
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DP-R212
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Canceled
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP-CTR212-III-03
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: DP-R212
MeSH Terms: conditions — Hypertension; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DP-R212 group (Experimental): DP-R212 + C1-R212 placebo + C2-R212 placebo
  Interventions: Drug: DP-R212
- C1-R212 group (Active Comparator): DP-R212 placebo + C1-R212 + C2-R212 placebo
  Interventions: Drug: C1-R212
- C2-R212 group (Active Comparator): DP-R212 placebo + C1-R212 placebo + C2-R212
  Interventions: Drug: C2-R212

INTERVENTIONS:
Drug: DP-R212 — DP-R212 + C1-R212 placebo + C2-R212 placebo
  Arms: DP-R212 group
Drug: C1-R212 — DP-R212 placebo + C1-R212 + C2-R212 placebo
  Arms: C1-R212 group
Drug: C2-R212 — DP-R212 placebo + C1-R212 placebo + C2-R212
  Arms: C2-R212 group

SUMMARY:
The purpose of this study is to determine superiority of DP-R212 comparing to each monotherapy in patient with hypertension and primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Both man and woman who is over 19 years old
* Hypertension patient with hypercholesterolemia

Exclusion Criteria:

* sSBP difference is ≥20mmHg or sDBP difference is ≥10mmHg
* A history of cardiovascular disease
* rhabdomyolysis, myopathy
* Hypertension or hypercholesterolemia due to secondary causes
* Uncontrolled diabetes
* Evidence of hepatic or renal disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Percent change of LDL-Cholesterol | 0, 8 weeks
Change of mean seated Systolic Blood Pressure | 0, 8 weeks

IPD SHARING:
Plan to Share IPD: No